CLINICAL TRIAL: NCT02778217
Title: The Blastocyst Development and Clinical Outcome in Single Step Medium With or Without Renewal on Day 3 in a Time-lapse Incubator
Brief Title: Blastocyst Culture in a Time-lapse Incubator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dar AlMaraa Center (Other)
Responsible Party: Principal Investigator, Yasmin, Senior clinical embryologist, Dar AlMaraa Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 006734
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Sub-optimal Culture Conditions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uninterrupted single embryo culture (No Intervention): The same single medium is used throughout the 5-6 days of culture with no replenishment on day 3.
- Interrupted single medium culture (Experimental): The single step medium is renewed on Day 3 of embryo culture.
  Interventions: Procedure: Culture media renwal

INTERVENTIONS:
Procedure: Culture media renwal
  Arms: Interrupted single medium culture

SUMMARY:
Culture media used to support development of zygotes to the blastocyst stage is based on two basic philosophies: a single step medium "let-the-embryo-choose" or a sequential medium "back-to-nature".

For single step media, there are two types of protocol can be used for the culture of human preimplantation embryos:

1. Interrupted single medium culture, in which the medium is renewed on the Day 3 of embryo culture
2. Uninterrupted single embryo culture, in which the same single medium is used throughout the 5-6 days of culture with no replenishment or replacement on Day 3.

Investigators aim to compare the blastocyst development and clinical outcome between the two types of protocols of a single medium (with or without renewal on Day 3)

ELIGIBILITY:
Inclusion Criteria:

* female partners were under the age of 39 years
* Intracytoplasmic sperm injection (ICSI) was performed using fresh ejaculates

Exclusion Criteria:

* Day 3 embryo transfer cycles

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks post embryo transfer
  diagnosed by the presence of a heartbeat in the gestational sac visualized by ultrasound

SECONDARY OUTCOMES:
Implantation rate | 4-6 weeks post embryo transfer
  the number of intrauterine gestational sacs over the total number of embryos transferred
Blastocyst formation rate | 5-6 days post intracytoplasmic sperm injection

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Magdi, M.Sc, Principal Investigator — Dar Almaraa fertility and gynacology center
Locations (1):
- Sunrise fertility center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Costa-Borges N, Belles M, Meseguer M, Galliano D, Ballesteros A, Calderon G. Blastocyst development in single medium with or without renewal on day 3: a prospective cohort study on sibling donor oocytes in a time-lapse incubator. Fertil Steril. 2016 Mar;105(3):707-713. doi: 10.1016/j.fertnstert.2015.11.038. Epub 2015 Dec 12. PMID 26690010